CLINICAL TRIAL: NCT03587818
Title: Person-Centred Information and Communication for Patients Undergoing Colo-Rectal Surgery - the PINCORE Project: a Quasi-experimental Longitudinal Design
Brief Title: Person-Centred Information and Communication for Patients Undergoing Colo-Rectal Surgery - the PINCORE Project
Acronym: PINCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: GPCC core project PINCORE
Record Dates: First submitted 2018-04-25; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Neoplasms
Keywords: Patient-Centered Care; Health Communication; Clinical trial; Colorectal neoplasms; Colorectal surgery; Continuity of patient care; Medical-surgical nursing; Qualitative Research
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A before and after design was performed; the control group were included from November 2012 to January 2014. This was followed by introducing the intervention to the clinicians, and the intervention group were included from March 2014 to June 2015. Patients were assigned consecutively at the three hospitals. No blinding was applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Conventional care. Patients were receiving several written patient education materials (PEMs), mostly related to specific parts or procedures related to the surgery and the recovery.
  Communication between patients and professionals during consultations occurred according to conventional care practice.
- Intervention group (Experimental): I. Written interactive PEM structured into chapters/phases of the care process. Designed to serve three purposes:
  1. generic information of the surgery and recovery process on a group level to promote high readability, suitability and comprehensibility
  2. arena of dialogues between patient and professionals; voicing concerns, share perspectives
  3. for the patient to personally reflect on generic information.
  II. Person-centred communication in dialogues using the PEM as a supportive tool, facilitated by four communication strategies:
  1. professionals guiding the patient through the care process
  2. communicating an introduction, agenda and closing
  3. being sensitive to the patient's questions, beliefs, experiences and resources
  4. dialogue based on story, posing open-ended questions, and following up.
  Interventions: Other: person-centred communication

INTERVENTIONS:
Other: person-centred communication — The intervention aimed to actively make use of a person-centred approach to support patients undergoing CRC surgery to be prepared for surgery, discharge and recovery in relation to CRC. This was accomplished through person-centred communication, which was based on a standardized dialogue tool with tailored written information material (component I), in combination with an approach for professionals to facilitate person-centred communication (component II) in consultations.
  Arms: Intervention group

SUMMARY:
An overarching aim is to create prerequisites for person-centred information and communication. The specific aim is to evaluate if an intervention with a written information and communication support tool and person-centred dialogues can increase patients' health-related quality of life and preparedness and well-being pre-surgery and during recovery in connection to colorectal cancer (CRC) surgery. Further, the aim is to explain variations in patients' recovery trajectories during the six months following CRC surgery in order to identify particularly vulnerable sub-groups of patients.

The hypothesis is that person-centred information and communication supported by an interactive patient information and education material (PEM) for patients undergoing CRC surgery will lead to improved preparedness for surgery and recovery during recovery 6 months following surgery. Secondary outcomes were decreased length of stay at hospital in relation to surgery, changed behaviour pertaining when and how to seek health care for recovery support, and improved emotional, role and social function, general health status and distress.

The study is performed at three surgical departments in Sweden. A combination of quantitative and qualitative methods will be applied. The project started with analysis of existing patient written information and education materials aimed for the patient group at Swedish surgical departments and analyses of conversations between patients and providers in consultations occurring over time before and following surgery. These results provided the basis for the development of the person-centred communication intervention developed in collaboration between people who had undergone CRC surgery, professionals from CRC surgery clinics and researchers with expertise in patient education, person-centred care and CRC surgery.

The design is quasi-experimental and longitudinal. Patients are consecutively sampled. Types of data:

* patient reported answers in validated questionnaires
* information about diagnosis, type of treatments and course of care obtained from patients' records
* recorded consultation conversations with patients between patients and health care providers
* narrative interviews with patients 6 months following discharge regarding their recovery after surgery
* focus group discussions and individual interviews with professionals regarding how they have perceived using the intervention and how it has functioned.

DETAILED DESCRIPTION:
Background In Sweden, approximately 3,900 people are diagnosed with colon cancer and 1,900 with rectal cancer annually, split almost equally between women and men. The primary treatment for colorectal cancer (CRC) is surgery. A particular challenge in CRC care is meeting patients' information needs over time in order to improve their recovery. There is a need for comprehensive considerations and person-centred communication supporting patients to be prepared for the surgery and the following recovery.

Aim An overarching aim is to create prerequisites for person-centred information and communication. The specific aim is to evaluate if an intervention with a written information and communication support tool and person-centred dialogues can increase patients' health-related quality of life and preparedness and well-being pre-surgery and during recovery in connection to colorectal cancer surgery. The hypothesis is that person-centred information and communication supported by an interactive patient information and education material (PEM) for patients undergoing CRC surgery will lead to improved preparedness for surgery and recovery during recovery 6 months following surgery. Secondary outcomes were decreased length of stay at hospital in relation to surgery, changed behaviour pertaining when and how to seek health care for recovery support, and improved emotional, role and social function, general health status and distress. Further, the aim is to explain variations in patients' recovery trajectories during the six months following CRC surgery in order to identify particularly vulnerable sub-groups of patients.

Communication in consultations will be supported by a innovative written interactive PEM with the goal to enhance the patient's knowledge seeking in order to be prepared for "the next step" in his/her care process. Here, person-centred communication refers to the patient-provider conversations where the patient is encouraged to tell about personal experiences, perceptions and worries in a dialogue format. An assumption is that dialogues unfolds when the two partners together are seeking to make sense of what is shared to each others.

Method Three hospitals. The study is performed at three surgical departments; university, regional and local hospitals; including public and private non-profit. Health care providers and patients from the three hospitals will be included in the development and evaluation of the intervention. A combination of quantitative and qualitative methods will be applied.

Initial analyses before the development of the intervention The project started with analysis of existing patient written information and education materials aimed for the patient group at Swedish surgical departments and analyses of conversations between patients and providers in consultations occurring over time before and following surgery. These results provided the basis for the development of the person-centred communication intervention developed in collaboration between people who had undergone CRC surgery, professionals from CRC surgery clinics and researchers with expertise in patient education, person-centred care and CRC surgery.

Evaluation in a quasi-experimental design

The design of the clinical intervention study is quasi-experimental and longitudinal; one group of patients before the introduction of the intervention will be compared to one group who have been part of the intervention (consecutively sampled). For the evaluation several types of data will be used:

* patient reported answers in validated questionnaires
* clinical and treatment data obtained from patients' records
* recorded consultation conversations with patients between patients and health care providers
* narrative interviews with patients 6 months following discharge regarding their recovery after surgery
* focus group discussions and individual interviews with professionals regarding how they have perceived using the intervention and how it has functioned

Expected result The project will contribute a model for the enabling of person-centred communication in connection to CRC surgery. There are many people who will benefit of improved support for the specific group of patients, since CRC is a common type of cancer affecting women and men and where surgery is the most common treatment. Evaluations with a combination of methods increase the possibility to explain the significance of the intervention and how it can be implemented. The design of the intervention model, including a video and workshop outline for the introduction of the intervention model to health care professionals, facilitates direct clinical implementation if the evaluation will be proved effective. The written interactive PEM developed and tested is general for the Swedish context and include a generic approach for how to design the interactive PEM to other groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* undergoing planned surgery for cancer in colon or rectum

Exclusion Criteria:

* receiving preoperative chemotherapy
* receiving long-term preoperative radiation
* diagnosed metastasis
* post-surgical diagnosis of benign tumors
* undergoing emergency surgery
* having reduced cognitive function
* lacking ability to communicate in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
The Longitudinal Preparedness for Colorectal Cancer Surgery Questionnaire (PCSQ) | six months after surgery
  measures change in preparedness for surgery and recovery over time in four domains: (i) searching for and making use of information (4 items), (ii) understanding and involvement in the care process (7 items), (iii) making sense of the recovery process (5 items), and (iv) support and access to medical care (7 items)

SECONDARY OUTCOMES:
EORTC QLQ-C30 version 3.0 | (1) before surgery, (2) six weeks after surgery, (3) three months after surgery and (4) six months after surgery
  Functional status scales measuring physical functioning (5 items), emotional functioning (4 items), role functioning (2 items), cognitive functioning (2 items) and social functioning (2 items) and global health status/QoL (2 items), and symptom scales for fatigue (3 items), nausea and vomiting (2 items), and pain (2 items), single items for dyspnoea, insomnia, appetite loss, constipation and diarrhoea, and financial difficulties.
The National Comprehensive Cancer Network (NCCS) Distress Thermometer (DT; Version 1.2013). | (1) before surgery, (2) one week after surgery, (3) six weeks after surgery, (4) three months after surgery and (5) six months after surgery
  A one item thermometer visual analogue scale, accompanied with a Problem list categorized into five subscales: practical (6 items), family (4 items), emotional (6 items), physical (22 items), and spiritual/religious (1 items).
The Daily Coping Assessment instrument | (1) one week after surgery and (2) six weeks after surgery.
  Number and types of pre-defined situational coping strategies used during the day to handle what the person perceives as the most stressful event, illness-related or not.
Communication in consultations | Pre-surgery
  Audio-recorded planned consultations between patients and professionals.
Patients experience of the recovery process | 6 months following surgery
  Audio-recorded individual narrative interviews with patients.
Orientation to Life Questionnaire (OLQ-13) | (1) before surgery and (2) six months after surgery
  13 items that measure sense of coherence on meaningfulness (4 items), manageability (4 items) and comprehensibility (5 items). Items are scored on 7-point scales.
Length of stay at hospital in relation to surgery | (1) before surgery and (2) within 6 months after surgery
  Days hospitalised; obtained from patients' medical records
Behaviour pertaining when and how to seek health care for recovery support: Telephone-calls | (1) before surgery and (2) within 6 months after surgery
  Numbers of calls; obtained from patients' medical records
Behaviour pertaining when and how to seek health care for recovery support: Visits at outpatients clinics | (1) before surgery and (2) within 6 months after surgery
  Numbers of visits; obtained from patients' medical records

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Öhlén, PhD, Principal Investigator — Göteborg University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Smith F, Carlsson E, Kokkinakis D, Forsberg M, Kodeda K, Sawatzky R, Friberg F, Ohlen J. Readability, suitability and comprehensibility in patient education materials for Swedish patients with colorectal cancer undergoing elective surgery: a mixed method design. Patient Educ Couns. 2014 Feb;94(2):202-9. doi: 10.1016/j.pec.2013.10.009. Epub 2013 Nov 5. PMID 24290242
- [Result] Oresland S, Friberg F, Maatta S, Ohlen J. Disclosing discourses: biomedical and hospitality discourses in patient education materials. Nurs Inq. 2015 Sep;22(3):240-8. doi: 10.1111/nin.12097. Epub 2015 Apr 6. PMID 25847051
- [Result] Carlsson E, Pettersson M, Hyden LC, Ohlen J, Friberg F. Structure and content in consultations with patients undergoing surgery for colorectal cancer. Eur J Oncol Nurs. 2013 Dec;17(6):820-6. doi: 10.1016/j.ejon.2013.07.002. Epub 2013 Sep 5. PMID 24012188
- [Result] Pettersson ME, Ohlen J, Friberg F, Hyden LC, Carlsson E. Topics and structure in preoperative nursing consultations with patients undergoing colorectal cancer surgery. Scand J Caring Sci. 2017 Dec;31(4):674-686. doi: 10.1111/scs.12378. Epub 2016 Nov 8. PMID 27859450
- [Result] Friberg F, Liden E, Hakanson C, Ohlen J. Communicating bodily changes: physicians' ways of enabling patient understanding in gastrointestinal cancer consultations. Palliat Support Care. 2015 Jun;13(3):661-71. doi: 10.1017/S1478951514000352. Epub 2014 May 2. PMID 24784141
- [Result] Carlsson E, Pettersson M, Ohlen J, Sawatzky R, Smith F, Friberg F. Development and validation of the preparedness for Colorectal Cancer Surgery Questionnaire: PCSQ-pre 24. Eur J Oncol Nurs. 2016 Dec;25:24-32. doi: 10.1016/j.ejon.2016.09.002. Epub 2016 Sep 21. PMID 27865249
- [Result] Sawatzky R, Russell L, Friberg F, Carlsson EK, Pettersson M, Ohlen J. Longitudinal person-centered measurement: A psychometric evaluation of the Preparedness for Colorectal Cancer Surgery Questionnaire (PCSQ). Patient Educ Couns. 2017 May;100(5):827-835. doi: 10.1016/j.pec.2016.11.010. Epub 2016 Nov 15. PMID 27955903
- [Result] Smith F, Ohlen J, Persson LO, Carlsson E. Daily Assessment of Stressful events and Coping in early post-operative recovery after colorectal cancer surgery. Eur J Cancer Care (Engl). 2018 Mar;27(2):e12829. doi: 10.1111/ecc.12829. Epub 2018 Jan 24. PMID 29363821
- [Result] Smith F, Wallengren Gustafsson C & Öhlén J. (2017) Participatory design in education materials in health care context. Action Research 15(3), 310-336.